CLINICAL TRIAL: NCT02688933
Title: A Randomized, Active-controlled, Parallel Group, 16-Week Open Label Study Comparing the Efficacy and Safety of the Morning Injection of Toujeo (Insulin Glargine-U300) Versus Lantus in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study Comparing the Efficacy and Safety of the Morning Injection of Toujeo Versus Lantus in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14587; U1111-1176-0936 (Other: UTN)
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE901-U300 (Experimental): HOE901-U300 (Insulin glargine, 300 U/mL) once daily for 16 weeks on top of mealtime insulins analogs. Basal insulin doses were individually titrated (until the end of Week 14) to reach fasting self-measured plasma glucose (SMPG) levels of 80 to 100 mg/dL, while mitigating hypoglycemia.
  Interventions: Drug: HOE901-U300 (Insulin Glargine 300 U/ml); Drug: Mandated back ground therapy
- Lantus (Active Comparator): Lantus (Insulin glargine, 100 U/mL) once daily for 16 weeks on top of mealtime insulins analogs. Basal insulin doses were individually titrated (until the end of Week 14) to reach fasting SMPG levels of 80 to 100 mg/dL, while mitigating hypoglycemia.
  Interventions: Drug: Lantus (Insulin Glargine 100 U/ml); Drug: Mandated back ground therapy

INTERVENTIONS:
Drug: HOE901-U300 (Insulin Glargine 300 U/ml) — Self-administered by subcutaneous (SC) injection in the morning (between waking up and breakfast) using a pre-filled pen.
  Other Names: Toujeo
  Arms: HOE901-U300
Drug: Lantus (Insulin Glargine 100 U/ml) — Self-administered by subcutaneous (SC) injection in the morning (between waking up and breakfast using a pre-filled pen.
  Other Names: HOE901-U100
  Arms: Lantus
Drug: Mandated back ground therapy — Rapid insulin analogs: e.g., insulin glulisine, insulin lispro or insulin aspart, used by participant at least 30 days before screening. Mealtime insulin was to be continued during the study and titrated towards protocol specified postprandial glucose targets (130-180 mg/dL).

SUMMARY:
Primary Objective:

To demonstrate that morning injection of Toujeo (HOE901-U300) compared to Lantus provides better glycemic control evaluated by Continuous Glucose Monitoring (CGM) in adult participants with type 1 diabetes mellitus.

Secondary Objective:

To demonstrate that treatment with HOE901-U300 compared to Lantus provides:

* Lower incidence rate of nocturnal symptomatic hypoglycemia;
* Better glucose control coverage during the last hours of CGM before next basal-insulin dosing;
* Less variability in CGM profile.

DETAILED DESCRIPTION:
The maximum study duration per participant was to be of approximately 20 weeks that consisted of an up to a 4-week screening and CGM training period including a 1-2 week baseline (blinded) CGM performance (allowed for re-training), a 14-week open-label, comparative treatment period allowing for dose titration in both basal and meal-time insulin and including a 1-2 week end-of treatment blinded CGM collection with fixed dose of HOE901-U300 and Lantus, and a 2 day post treatment follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Adult participants (male and female) with type 1 diabetes mellitus (T1DM).
* Signed written informed consent.

Exclusion criteria:

* Age <18 years or >70 years.
* Fasting c-peptide ≥0.3 nmol/L as per source document or central lab test at Visit 1.
* Glycated hemoglobin (HbA1c) ≤ 6.5 % or ≥ 10.0% via central lab test at Visit 1.
* Participants who experienced none of episode of documented symptomatic and/or severe hypoglycemia (as per the American Diabetes Association (ADA) classification) during the past month prior to screening.
* Participants who experienced >1 episode of severe hypoglycemia resulting in coma/seizures during the last 12 months before screening.
* Participants received less than 1 year treatment with basal plus mealtime insulin.
* Used any basal insulins other than long-acting insulin analogs (ie, Lantus, Toujeo, Levemir, and Tresiba) in the past 3 months before screening.
* Required >80 U/day basal insulin analogs or not on stable dose (±20% total dose) within 30 days prior to screening.
* Used fewer than 2 injections of rapid-acting insulin analog per day within 30 days prior to screening.
* Used human regular insulin as mealtime insulin within 30 days prior to screening.
* Used an insulin pump during the last 6 months before screening.
* History of unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to required treatment (e.g., laser, surgical treatment, or injectable drugs) during the study period.
* Pregnant or breast-feeding women or planned pregnancy during the duration of the study.
* Use of any other investigational drug(s) within 1 month or 5 half-lives, whichever was longer prior to screening.
* Inappropriate CGM use during screening period evidenced by failure to obtain a minimum of 4 days of usable records by the end of screening.
* Noncompliance with self-monitored plasma glucose (SMPG) performance evidenced by failure to demonstrate at least 5 days of 5 point SMPG records by the end of screening.

The above information is not intended to contain all considerations relevant to a participants's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (100):
- United States (99):
  - Investigational Site Number 840-151, Little Rock, Arkansas
  - Investigational Site Number 840-071, Concord, California
  - Investigational Site Number 840-149, Escondido, California
  - Investigational Site Number 840-004, Fresno, California
  - Investigational Site Number 840-110, Greenbrae, California
  - Investigational Site Number 840-124, La Jolla, California
  - Investigational Site Number 840-030, La Mesa, California
  - Investigational Site Number 840-044, Los Angeles, California
  - Investigational Site Number 840-022, Los Angeles, California
  - Investigational Site Number 840-129, Los Gatos, California
  - Investigational Site Number 840-024, Northridge, California
  - Investigational Site Number 840-069, Pomona, California
  - Investigational Site Number 840-090, Pomona, California
  - Investigational Site Number 840-132, Rolling Hills Estates, California
  - Investigational Site Number 840-130, San Jose, California
  - Investigational Site Number 840-055, San Ramon, California
  - Investigational Site Number 840-028, Santa Barbara, California
  - Investigational Site Number 840-063, Tarzana, California
  - Investigational Site Number 840-138, Tustin, California
  - Investigational Site Number 840-016, Ventura, California
  - Investigational Site Number 840-039, Denver, Colorado
  - Investigational Site Number 840-021, Denver, Colorado
  - Investigational Site Number 840-070, Denver, Colorado
  - Investigational Site Number 840-046, Englewood, Colorado
  - Investigational Site Number 840-072, Coral Gables, Florida
  - Investigational Site Number 840-133, Hialeah, Florida
  - Investigational Site Number 840-137, Maitland, Florida
  - Investigational Site Number 840-049, Miami, Florida
  - Investigational Site Number 840-076, Miami, Florida
  - Investigational Site Number 840-023, New Port Richey, Florida
  - Investigational Site Number 840-053, Ocoee, Florida
  - Investigational Site Number 840-112, Ormond Beach, Florida
  - Investigational Site Number 840-018, Palm Harbor, Florida
  - Investigational Site Number 840-047, Port Charlotte, Florida
  - Investigational Site Number 840-114, Tampa, Florida
  - Investigational Site Number 840-036, West Palm Beach, Florida
  - Investigational Site Number 840-001, Atlanta, Georgia
  - Investigational Site Number 840-064, Columbus, Georgia
  - Investigational Site Number 840-012, Lawrenceville, Georgia
  - Investigational Site Number 840-008, Roswell, Georgia
  - Investigational Site Number 840-014, Stockbridge, Georgia
  - Investigational Site Number 840-060, Idaho Falls, Idaho
  - Investigational Site Number 840-125, Arlington Heights, Illinois
  - Investigational Site Number 840-011, Chicago, Illinois
  - Investigational Site Number 840-134, Crystal Lake, Illinois
  - Investigational Site Number 840-002, West Des Moines, Iowa
  - Investigational Site Number 840-073, Wichita, Kansas
  - Investigational Site Number 840-062, Covington, Kentucky
  - Investigational Site Number 840-042, Lexington, Kentucky
  - Investigational Site Number 840-009, Metairie, Louisiana
  - Investigational Site Number 840-032, New Orleans, Louisiana
  - Investigational Site Number 840-054, Hyattsville, Maryland
  - Investigational Site Number 840-006, Rockville, Maryland
  - Investigational Site Number 840-157, Framingham, Massachusetts
  - Investigational Site Number 840-122, Waltham, Massachusetts
  - Investigational Site Number 840-037, Flint, Michigan
  - Investigational Site Number 840-067, Billings, Montana
  - Investigational Site Number 840-094, Lincoln, Nebraska
  - Investigational Site Number 840-033, Omaha, Nebraska
  - Investigational Site Number 840-142, Omaha, Nebraska
  - Investigational Site Number 840-040, Henderson, Nevada
  - Investigational Site Number 840-017, Las Vegas, Nevada
  - Investigational Site Number 840-102, New York, New York
  - Investigational Site Number 840-108, New York, New York
  - Investigational Site Number 840-109, Staten Island, New York
  - Investigational Site Number 840-045, Greenville, North Carolina
  - Investigational Site Number 840-010, Morehead City, North Carolina
  - Investigational Site Number 840-080, Morehead City, North Carolina
  - Investigational Site Number 840-051, Fargo, North Dakota
  - Investigational Site Number 840-123, Columbus, Ohio
  - Investigational Site Number 840-104, Mentor, Ohio
  - Investigational Site Number 840-079, Norman, Oklahoma
  - Investigational Site Number 840-162, Bend, Oregon
  - Investigational Site Number 840-096, Portland, Oregon
  - Investigational Site Number 840-058, Chattanooga, Tennessee
  - Investigational Site Number 840-003, Dallas, Texas
  - Investigational Site Number 840-019, Dallas, Texas
  - Investigational Site Number 840-075, Dallas, Texas
  - Investigational Site Number 840-005, Dallas, Texas
  - Investigational Site Number 840-013, Dallas, Texas
  - Investigational Site Number 840-153, El Paso, Texas
  - Investigational Site Number 840-026, Fort Worth, Texas
  - Investigational Site Number 840-081, Houston, Texas
  - Investigational Site Number 840-160, Houston, Texas
  - Investigational Site Number 840-156, Houston, Texas
  - Investigational Site Number 840-152, Houston, Texas
  - Investigational Site Number 840-031, Houston, Texas
  - Investigational Site Number 840-140, Lufkin, Texas
  - Investigational Site Number 840-029, Mesquite, Texas
  - Investigational Site Number 840-048, North Richland Hills, Texas
  - Investigational Site Number 840-150, Pearland, Texas
  - Investigational Site Number 840-083, Murray, Utah
  - Investigational Site Number 840-101, Ogden, Utah
  - Investigational Site Number 840-097, Salt Lake City, Utah
  - Investigational Site Number 840-143, Bennington, Vermont
  - Investigational Site Number 840-056, Burlington, Vermont
  - Investigational Site Number 840-015, Renton, Washington
  - Investigational Site Number 840-074, Spokane, Washington
  - Investigational Site Number 840-139, Bridgeport, West Virginia
- Investigational Site Number 840-111, Manatí, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 100 sites in United States. A total of 980 participants were screened between 5 May 2016 and 16 February 2017, of whom 342 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: A total of 638 participants were randomized in HOE901-U300 or Lantus, stratified by baseline HbA1c (<8 %,> =8%), frequency of basal insulin injections at Visit 1 (twice vs once daily), current continuous glucose monitoring (CGM) use at Visit 1(yes/no) and mealtime insulin titration algorithm (simple titration vs carbohydrate counting).
Groups:
- HOE901-U300: HOE901-U300 (Insulin glargine, 300 U/mL) subcutaneous (SC) injection once daily up to Week 16 on top of mealtime insulin analogs. Basal insulin doses were individually titrated to reach fasting self-measured plasma glucose (SMPG) levels within the target range of 80 to 100 mg/dL.
- Lantus: Lantus (Insulin glargine, 100 U/mL) SC injection once daily up to Week 16 on top of mealtime insulin analogs. Basal insulin doses were individually titrated to reach fasting SMPG levels within the target range of 80 to 100 mg/dL.
Period: Overall Study
Arm/Group | HOE901-U300 | Lantus
Started | 320 | 318
Completed | 291 | 281
Not Completed | 29 | 37
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 2 | 2
Not completed — Poor compliance to protocol | 7 | 4
Not completed — Hypoglycemia | 2 | 0
Not completed — Other than Specified | 14 | 25
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population that included any participant who had been allocated to a randomized treatment regardless of whether the treatment kit was used or not.
Groups:
- HOE901-U300: HOE901-U300 (Insulin glargine, 300 U/mL) SC injection once daily up to Week 16 on top of mealtime insulin analogs. Basal insulin doses were individually titrated to reach fasting SMPG levels within the target range of 80 to 100 mg/dL.
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 | Lantus | Total
Number analyzed (Participants) | 320 | 318 | 638
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (14.0) | 45.5 (13.9) | 45.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 138 | 278
  Male | 180 | 180 | 360
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 42 | 85
  Not Hispanic or Latino | 277 | 276 | 553
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 24 | 28 | 52
  White | 281 | 282 | 563
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 4 | 10
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.50 (4.88) | 27.65 (4.92) | 27.57 (4.90)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time of Mean Glucose Concentration Within the Target Range of 70-180 mg/dL as Obtained From CGM
Description: The CGM system combined frequent interstitial glucose measurements (every 5 minutes) with ability to analyze glucose levels in real time. Adjusted least square (LS) means and standard error (SE) were obtained from a generalized linear model with identity link including post baseline CGM assessment during Week 15 (and/or Week 16).
Time Frame: During Week 15 and/or 16
Population: Modified intent-to-treat (mITT) population that included all participants who were randomized and had a post-baseline CGM assessment and enough CGM data values to calculate the primary outcome measure, percent of time in range of 70-180 mg/dL during Week 15 (and/or Week 16).
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
percentage of time | 55.40 (1.08) | 55.18 (1.10)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was performed using generalized linear model with identity link, had percentage of time glucose concentration within target range 70-180 mg/dL as dependent variable, treatment group as an independent variable, adjusting variables including baseline characteristics: duration of diabetes, baseline BMI, age, and randomization strata (HbA1c at screening [<8.0% vs ≥8.0%], frequency of Lantus injection at screening, current CGM use [yes/no], and mealtime insulin titration algorithm); Test type: Superiority; p = 0.8494, Generalized linear model — Threshold for significance at 0.05 level; Generalized linear model with identity link; Least Square mean difference = 0.22, Standard Error of Mean 1.15

2. Secondary Outcome: Percentage of Participants With Documented Symptomatic Nocturnal Hypoglycemia
Description: Documented symptomatic nocturnal hypoglycemia was defined as an event with typical symptoms of hypoglycemia accompanied by SMPG <=70 mg/dL that occurred between 00:00 and 05:59 hours as reported on the hypoglycemia electronic case report form (eCRF).
Time Frame: Baseline up to Week 16
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
percentage of participants
  Documented <=70mg/dL | 70.8 | 68.3
  Documented <54 mg/dL | 50.9 | 54.1

3. Secondary Outcome: Documented Symptomatic Nocturnal Hypoglycemia Event Rate Per Participant-Year
Description: Documented symptomatic nocturnal hypoglycemia was defined as an event with typical symptoms of hypoglycemia accompanied by SMPG <=70 mg/dL that occurred between 00:00 and 05:59 hours as reported on the hypoglycemia eCRF.
Time Frame: Baseline up to Week 16
Population: mITT population.
Measure: Number; unit: events per participant-year
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
events per participant-year
  Documented <=70 mg/dL | 11.38 | 11.39
  Documented <54 mg/dL | 4.99 | 5.61

4. Secondary Outcome: Mean Change From Baseline in Glucose Level During Last 4 Hours of CGM Data Collection Prior to the Next Day Basal Insulin Injection During Week 15 and/or Week 16
Description: Adjusted LS means and SE were obtained from mixed model including post baseline CGM assessment during the last 4 hours prior to the next day's basal insulin injection during Week 15 (and/or Week 16).
Time Frame: Baseline, during Week 15 and/or Week 16
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
mg/dL | -1.99 (3.68) | 5.67 (3.72)

5. Secondary Outcome: Percentage of Time Glucose Concentrations Within the Target Range of 70 to 140 mg/dL During Last 4 Hours of CGM Data Collection Prior to Next Day Basal Insulin Injection
Description: as for outcome 4
Time Frame: During Week 15 and/or Week 16
Population: mITT population
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
percentage of time | 36.49 (1.62) | 35.07 (1.65)

6. Secondary Outcome: Coefficient of Variation (CV%) in Mean CGM Glucose
Description: CV% was a measure of spread of variability relative to mean of population. For CGM glucose values over 24 hours, CV% was measure of glycemic variability across 24-hour day and calculated for each period (total, within day and between days) as ratio of standard deviation of glucose values to mean of glucose values.
Time Frame: During Week 15 and/or Week 16
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent of mean glucose level
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
percent of mean glucose level
  Total CV% | 41.27 (0.63) | 40.72 (0.64)
  Within-day CV% | 36.99 (0.56) | 36.23 (0.56)
  Between-days CV% | 17.44 (0.59) | 17.53 (0.60)

7. Other Pre Specified Outcome: Change From Baseline in Daily Insulin Dose at Week 16
Description: Change from Baseline at Week 16 for daily basal insulin dose and daily bolus insulin dose was reported.
Time Frame: Baseline, Week 16
Population: Safety population: all participants who took at least 1 dose of randomized treatment & analyzed as-treated (as per treatment actually received) also to whom it was unclear whether they took study medication & who received more than 1 study treatment during trial. Here, "number analyzed": number of participants evaluable for each specified category.
Measure: Mean (Standard Deviation); unit: International Units
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 320 | 318
International Units
  Daily basal Insulin Dose: number analyzed (Participants) | 295 | 283
  Daily basal Insulin Dose | 8.8 (11.8) | 7.0 (10.1)
  Daily bolus Insulin Dose: number analyzed (Participants) | 218 | 209
  Daily bolus Insulin Dose | -1.8 (11.8) | -3.0 (11.3)

8. Post Hoc Outcome: Change From Baseline in Time (Min) of Mean Glucose Concentration Within the Target Range of 70 to 180 mg/dL, by End of Study hbA1c Levels During Week 15 and/or Week 16
Description: Adjusted LS means and SE were obtained from mixed model including post baseline CGM assessments. Data was reported for participants with an end of study HbA1c <7.5 or HbA1c >=7.5% over a 24 hour period.
Time Frame: Baseline, during Week 15 and/or Week 16
Population: mITT population. Here, "number analyzed" signifies the number of participants evaluable for each specified category.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 277 | 268
minutes
  End of study HbA1c <7.5%: number analyzed (Participants) | 136 | 146
  End of study HbA1c <7.5% | 105.84 (25.64) | 56.07 (25.40)
  End of study HbA1c >=7.5%: number analyzed (Participants) | 118 | 107
  End of study HbA1c >=7.5% | 11.64 (27.26) | 31.95 (27.57)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of informed consent form up to study completion (Week 16) regardless of seriousness or relationship to study drug.
Description: Reported AEs are treatment-emergent AEs developed/worsened during on treatment period (time from first dose of investigational medicinal product [IMP] up to one day after last dose of IMP).
Arm/Group | HOE901-U300 | Lantus
All-Cause Mortality (participants affected / at risk) | 0/320 | 0/318
Serious Adverse Events (participants affected / at risk) | 17/320 | 14/318
Other Adverse Events (participants affected / at risk) | 54/320 | 54/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=320) | Lantus (N=318)
Diabetic foot infection (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3
Depression (Psychiatric disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 0 | 1
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 2 | 3
Hypoglycaemic unconsciousness (Nervous system disorders) | 6 | 3
Angle closure glaucoma (Eye disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Renal injury (Renal and urinary disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=320) | Lantus (N=318)
Nasopharyngitis (Infections and infestations) | 27 | 27
Upper respiratory tract infection (Infections and infestations) | 28 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT02688933/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT02688933/SAP_001.pdf